CLINICAL TRIAL: NCT06409975
Title: Evaluating the Feasibility and Acceptability of Mindful Self-Compassion Among Transgender and Nonbinary Young Adults
Brief Title: Feasibility and Acceptability of Mindful Self-Compassion Among Transgender and Nonbinary Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rhode Island (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2106682-1; 1K01AT012495-01 (NIH)
Record Dates: First submitted 2023-11-15; First posted 2024-05-10 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Healthy
Keywords: transgender; nonbinary; mindful self-compassion; feasibility; acceptability

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindful Self-Compassion Intervention (Experimental): All enrolled participants will complete the remotely delivered 8 week MSC intervention (described in interventions). Participants are encouraged to practice the formal meditations and/or informal skills taught each week between sessions. Participants will give feedback on self-compassion activities and the overall intervention. They will also complete several measures before, during, and after the intervention and at 3-month follow-up.
  Interventions: Behavioral: Mindful Self-Compassion (MSC)

INTERVENTIONS:
Behavioral: Mindful Self-Compassion (MSC) — MSC is an 8-week virtual intervention with weekly 2.5-hour sessions and a 4-hour retreat (between sessions 5 and 6) which will take place online via HIPAA-compliant Zoom. Each weekly session includes an opening meditation, reflection on weekly practice, short teaching, a weekly core meditation or informal practice discussion, short break, brief centering practice, weekly core reflective activity and discussion, and self compassion skill of the week practice. The 4-hour retreat is focused on engaging with the formal practices that have been taught in weeks 1-5.

SUMMARY:
The goal of this single-arm feasibility study is to evaluate the feasibility and acceptability of an 8-week mindful self-compassion intervention and associated data-collection plan among transgender and nonbinary young adults. Participants will be asked to:

* Complete weekly 2.5-hour virtual classes for 8 weeks and a 4-hour virtual retreat
* Practice specific activities in between classes for 20-30 minutes a day
* Answer survey questions before starting the intervention, half-way through the intervention, after the intervention, and 3-months after the intervention ends.

DETAILED DESCRIPTION:
The specific aims of this study are to: 1) evaluate the feasibility and acceptability of an 8-week Mindful Self-Compassion (MSC) intervention and data collection plan (pre-, post-, 3-month follow-up) with 5 consecutive groups of transgender and nonbinary young adults (TNYA), 2) evaluate the usability of MSC intervention activities by TNYA and determine whether MSC activities need to be tailored for TNYA, and 3) explore data collected throughout each intervention implementation to evaluate patterns of missingness and potential participant burden, intervention adherence, and reasons for dropout.

ELIGIBILITY:
Inclusion Criteria:

* transgender, nonbinary, genderqueer (or another non-cisgender identity)
* have reliable access to a smart phone or computer/tablet and the Internet and is reasonably able to make the time commitment required of the program (self-report)
* speak and understand English

Exclusion Criteria:

* has had formal mindfulness training (i.e. mindfulness-based stress reduction course) or engages in regular mindfulness practice (15 minutes more than twice a week for the last six months or more)
* Score 15 or higher on the patient health questionnaire-8 (PHQ-8)
* Score 2 or higher on the Columbia Suicide Severity Rating Scale
* Experienced an acute physical health crisis (e.g., chemotherapy, recovery from severe injury) (Germer & Neff, 2019, p. 80) in the past year
* Head trauma, seizure, or loss of consciousness in the past 6 months
* Reports a history of trauma AND Scores 14 or higher on Post-Traumatic Checklist, 6-item Civilian version
* Reports a diagnosis of a personality disorder
* Reports a diagnosis of schizophrenia or a history of psychosis
* Reports acute panic attack in the past month and history of acute panic attacks with concern/worry about having another one in the future OR Reports severe social anxiety which would make attending class too difficult
* Reports an acute episode of psychosis or suicide attempt in the past 12 months
* Has engaged in non-suicidal self-injury in the past 6 months
* Currently prescribed antipsychotic medications, benzodiazepine (equivalent to 30mg diazepam/day) or opioids (>40mg morphine equivalent/day)
* Prescribed any other psychiatric medication, including medication for opioid use disorder, whose dose has been changed in the past 8 weeks or is anticipated to change in the next 2 months.
* Currently engage in harmful drinking (5 or more drinks on one occasion (Flentje et al., 2020) more than once in the past 2 weeks; OR have any concerns about the expectation to not be using substances during group sessions
* has undergone detoxification from alcohol or other drugs and has been in sustained remission (with or without medication) for less than 1 year
* Has been hospitalized overnight for mental health related reasons in the past year (any diagnoses except bipolar disorder) OR have a diagnosis of bipolar disorder and have had an episode of mania or have been hospitalized in the past 2 years
* Reports any other acute physical or mental illness symptoms that may make group participation difficult

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — have a gender identity that is transgender, non-binary, genderqueer (i.e. not cisgender)
Enrollment: 50 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment of participants into study | immediately after the intervention
  Intervention feasibility will be determined by the ability to recruit adequate study samples (N=10 per cohort; 5 cohorts total)
Percent of Sample Completing the Intervention | immediately after the intervention
  Intervention feasibility will also be determined by the percent of participants who complete the intervention, defined as completing at least 6/8 intervention sessions.
Percent of participants who report satisfaction with MSC as Excellent or Good | immediately after the intervention, at 12-week follow-up
  Participant quantitative ratings (Excellent, Good, Fair, Poor, Awful) of their satisfaction with the intervention and qualitative feedback on intervention will be collected at the end of the intervention to evaluate the acceptability of the overall 8-week intervention and again at 12-week follow-up.
Likelihood of recommending to others | immediately after the intervention, at 12-week follow-up
  Participants will also be asked how likely they would be to recommend the intervention to others (0-not at all likely; 10-very likely) and the strongest reason for their rating [Net Promoter Score] at the end of the intervention and again at 12-week follow-up
Intent to use specific intervention activities in the future | immediately after the intervention
  Participant quantitative ratings (0 not useful -10 very useful) and qualitative feedback on formal meditations and informal practices will be collected at the end of the intervention to evaluate the usability of intervention/components, including the likelihood (0 not likely, 10- very likely) that they will use each activity in the future.
Percent of completed data at each data-collection point | baseline, intervention week 4, immediately after the intervention, and 12 weeks after the intervention is completed
  Percent of completed data collected at each time point (pre-intervention, mid-intervention, post-intervention, and 3-month follow-up) and the amount of time it takes to complete individual measures and all measures will be used to evaluate the feasibility of the data collection plan

SECONDARY OUTCOMES:
Frequency of Use of Intervention Activities and perceived usefulness | 12 weeks after the intervention is completed
  Participant quantitative ratings on the usefulness of each formal meditation and informal practice (0 not useful -10 very useful), frequency of use since the intervention ended (more than once a day, daily, a few times a week, weekly, a few times a month, monthly, once or twice since the intervention ended, not at all) as well qualitative feedback about how the activities have been incorporated in everyday life.
Percent of sample retained at follow-up | 12 weeks after the intervention is completed
  Total number of participants who complete the follow-up measures at 12 weeks divided by the number of participants who completed the intervention.

OTHER OUTCOMES:
Total Practice Time During Intervention Weeks | immediately after the intervention
  Total time spent will be calculated by summing participants' weekly self-reports of frequency (# days, 0-7) and duration of home practice (0-30+ minutes; 5 minute increments) with formal and informal self-compassion activities.

CONTACTS AND LOCATIONS:
Overall Officials: Jordon D Bosse, PhD, Principal Investigator — University of Rhode Island
Locations (1):
- N/A-- All study activities being conducted virtually, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Only demographic and quantitative data will be stored and preserved in Zenodo, an open dissemination research data repository. Only fully de-identified data will be shared with outside investigators at any time.
  Data dictionaries, codebooks, notes about required variable transformations for descriptive analyses (if needed), and the online survey will be created, shared, and associated with the relevant datasets. Each variable in the codebook will include a brief description of the item along with the question number and question text from the online survey, variable name, variable label, value labels, and standard codes for missing values. Descriptions of composite variables, if created, will also be provided. Data collection instruments will be provided in portable document format (PDF) whenever possible. If a data collection instrument cannot be shared directly due to copyright or other issues, a link to the source of the instrument will be provided.
Supporting Information: ICF, CSR
Time Frame: Data will be made within one year of completion of the grant activities or at the time of publication of a completed data analysis (whichever comes first).
Access Criteria: Researchers will be required to submit a request for data access through Zenodo, which will undergo scientific and community advisory board review to ensure scientific quality, relevance, feasibility, and adherence to best practices to the ethical conduct of research involving transgender and gender diverse persons.
  Upon request approval, a data use agreement will be signed by the researcher and, if relevant, their respective institutional official. Once the DUA has been fully executed and proof of IRB approval or exemption has been provided, approval will be granted in Zenodo and the researcher will receive a unique link to access the relevant data and other files.
  In view of the specificity of the project, interested investigators- particularly those who do not have members of the transgender community on their team- will be encouraged to form a collaborative arrangement with the study's investigators rather than simply receive the resources themselves.